CLINICAL TRIAL: NCT03876041
Title: Evaluation of Corticosteroid as Modulators of Humeral and Cellular Immune Response in Open Heart Surgery in Egyptian Population
Brief Title: Evaluation of Corticosteroid in Systemic Inflammatory Response Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa fawzy, principal investegator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ASSUITUU
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: SIRS; MiRNA-155; Treg
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Methylprednisolone Hemisuccinate; Methylprednisolone; dexamethasone 21-phosphate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexamethasone group (Active Comparator): this group will receive Dexamethasone: 0.1 to 0.3 mg/kg as single intra-operative dose and blood samples will be obtained from central venous blood at following time points: immediately after insertion during anesthetic induction (T1), 48hrs post-operative (T2), 72hrs post-operative (T3).
  Interventions: Drug: Dexamethasone phosphate
- methylprednisolone group (Active Comparator): this group will receive Methylprednisolone: 5-10mg/kg as single intra-operative dose and blood samples will be obtained from central venous blood at following time points: immediately after insertion during anesthetic induction (T1), 48hrs post-operative (T2), 72hrs post-operative (T3).
  Interventions: Drug: solumedrol

INTERVENTIONS:
Drug: solumedrol — intravenous solution for injection
  Other Names: methylprednisolone
  Arms: methylprednisolone group
Drug: Dexamethasone phosphate — intravenous solution for injection
  Other Names: dexamethasone
  Arms: dexamethasone group

SUMMARY:
Cardiac surgery and cardiopulmonary bypass (CPB) initiate a whole-body systemic inflammatory response (SIRS) characterized by the activation of leukocytes, monocytes, and the complement cascade. Multiple mediators of the inflammatory process are released, including cytokines, endothelin, adhesion molecules, and oxygen free radicals. An exaggerated release of these mediators may contribute to numerous postoperative end-organ complications, including myocardial dysfunction, neurologic impairment, respiratory failure, altered renal and hepatic function, bleeding disorders, and multiple organ failure. Although most cardiac surgical patients do not experience major adverse events, it is likely that the inflammatory response impairs clinical recovery to some degree in all patients.

A large number of therapeutic strategies have been developed to attenuate the inflammatory reaction to CPB and thereby enhance recovery of the cardiac surgical patient. Intraoperative corticosteroid administration has been studied extensively as a primary pharmacologic anti-inflammatory treatment option.

DETAILED DESCRIPTION:
Investigations have shown that clinical outcomes have been improved, worsened, or unaffected by the intraoperative administration of dexamethasone or methylprednisolone Limited data suggest that low-dose corticosteroids may be as effective as high-dose treatment in reducing complications but with fewer potential side effects MicroRNAs (miRNAs) are protein regulators that play an important role in a wide range of cellular functions. There is increasing evidence for the close relationship between miRNA expression, Th17 cell differentiation and disease pathology The miRNA, miR-155, which was the subject of this study, has a range of known biological functions, which include the induction of Toll like receptor (TLR) activation in monocytes /macrophages and the modulation of TLR signaling, facilitating pro-inflammatory cellular responses and initiating systemic inflammatory responses, as well as regulating Treg cell differentiation, maintenance, and function. The expression of this miRNA can be induced by inflammatory cytokines, such as tumor necrosis factor α (TNFα), that are released into the circulation in the initial stages of a systemic inflammatory response. In another study, demonstrated that miR-155 enhanced Treg and Th17 cell differentiation and Th17 cell function by targeting (suppressor of cytokine signaling 1) SOCS1.

In this study, the investigators will compare effect of low dose intra-operative corticosteroid (dexamethasone and methylprednisolone) as anti-inflammatory modulators through detection of T regulatory cells(Tregs) and IL-17 and correlate relation between Treg, IL-17 and micro RNA-155.

ELIGIBILITY:
Inclusion Criteria:

* open heart surgery with Cardiopulmonary bypass machine with relatively long bypass time more than 60 minute
* All patients Included in study with normal heart function

Exclusion Criteria:

* Left ventricular ejection fraction less than 40%
* acute infection such as sepsis or pneumonia, hepatic and renal failure, cancer or any autoimmune disease
* the use of steroid within 2 week prior to operation
* coagulation abnormalities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
measure anti-inflammatory effect through detection T regulatory cell level by4 color flow cytometry analysis to quantify % of Tregs (CD4, CD25,FoxP3) | 72 hours post operative
  in blood of all subjects
detect microRNA-155 | 72 hours post operative
  micro-RNA 155 is measured by RT-PCR

SECONDARY OUTCOMES:
measure pro-inflammatory cytokines | 72 hours post operative
  pro-inflammatory cytokines such as IL-1 and IL-6 by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa F Fathy, researcher, Principal Investigator — Assuit Medical school
Locations (1):
- Assuit university hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cicarelli DD, Bensenor FE, Vieira JE. Effects of single dose of dexamethasone on patients with systemic inflammatory response. Sao Paulo Med J. 2006 Mar 2;124(2):90-5. doi: 10.1590/s1516-31802006000200008. PMID 16878192
- [Background] Wang D, Tang M, Zong P, Liu H, Zhang T, Liu Y, Zhao Y. MiRNA-155 Regulates the Th17/Treg Ratio by Targeting SOCS1 in Severe Acute Pancreatitis. Front Physiol. 2018 Jun 8;9:686. doi: 10.3389/fphys.2018.00686. eCollection 2018. PMID 29937734
- [Background] Bocsi J, Hanzka MC, Osmancik P, Hambsch J, Dahnert I, Sack U, Bellinghausen W, Schneider P, Janousek J, Kostelka M, Tarnok A. Modulation of the cellular and humoral immune response to pediatric open heart surgery by methylprednisolone. Cytometry B Clin Cytom. 2011 Jul-Aug;80(4):212-20. doi: 10.1002/cyto.b.20587. Epub 2011 Mar 4. PMID 21374796
- [Background] Schadenberg AW, Vastert SJ, Evens FC, Kuis W, van Vught AJ, Jansen NJ, Prakken BJ. FOXP3+ CD4+ Tregs lose suppressive potential but remain anergic during transient inflammation in human. Eur J Immunol. 2011 Apr;41(4):1132-42. doi: 10.1002/eji.201040363. Epub 2011 Mar 7. PMID 21381018
- [Background] Soltani G, Abbasi Tashnizi M, Moeinipour AA, Ganjifard M, Esfahanizadeh J, Sepehri Shamloo A, Purafzali Firuzabadi SJ, Zirak N. Comparing the effect of preoperative administration of methylprednisolone and its administration before and during surgery on the clinical outcome in pediatric open heart surgeries. Iran Red Crescent Med J. 2013 Jun;15(6):483-7. doi: 10.5812/ircmj.8105. Epub 2013 Jun 5. PMID 24349746